CLINICAL TRIAL: NCT06057441
Title: Auditory and Visual Noise as Possible Non-pharmacological Treatment of ADHD in School Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: Lund University (Other)
Responsible Party: Principal Investigator, Emma Claesdotter-Knutsson, Associate Professor, Region Skane
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2023-02476-01
Record Dates: First submitted 2023-09-12; First posted 2023-09-28 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Attention Deficit Hyperactivity Disorder; Neurodevelopmental Disorders
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity; Neurodevelopmental Disorders

STUDY DESIGN:
Intervention Model Description: Patients will be recruited from Child and Adolescent Psychiatry in Lund. Typically developing children (TDC) will be recruited from schools.
  All participants will perform a cross over control study. Participants will perform the entire test battery at one occasion, containing no noise, auditory white noise and visual white pixel noise (two levels). Participants in the ADHD group will perform the tests unmedicated. The order of the noise stimulation and no noise, as well as the order of the tasks, will be randomized over participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- No noise stimulation (No Intervention): A prolonged fixation (PF) task and memory guided saccade (MGS) task will be performed without noise.
- Auditory white noise stimulation (Active Comparator): A prolonged fixation (PF) task and memory guided saccade (MGS) task will be performed in auditory white noise.
  Interventions: Device: Auditory noise stimulation
- Visual white pixel noise, 25% (Active Comparator): A prolonged fixation (PF) task and memory guided saccade (MGS) task will be performed in visual white pixel noise at 25%.
  Interventions: Device: Visual noise stimulation
- Visual white pixel noise, 50% (Active Comparator): A prolonged fixation (PF) task and memory guided saccade (MGS) task will be performed in visual white pixel noise at 50%.
  Interventions: Device: Visual noise stimulation

INTERVENTIONS:
Device: Auditory noise stimulation — Auditory white noise stimulation delivered at 78dB through earphones
  Arms: Auditory white noise stimulation
Device: Visual noise stimulation — Visual white pixel noise stimulation, backgound pixel noise visible at computer screen
  Arms: Visual white pixel noise, 25%; Visual white pixel noise, 50%

SUMMARY:
The goal of this study is to compare the influence of visual and auditory white noise on performance in children with attention deficit hyperactivity disorder (ADHD). The main questions it aims to answer are:

* Can auditory white noise stimulation affect cognitive performance?
* Can visual white pixel noise affect cognitive performance? Participants will complete two eye tracking tasks under different sensory noise stimulation.

Researchers will compare the ADHD group with a group of typically developing children to see if the noise influences the groups differently and if it has the potential to affect the performance of the ADHD group, to reach the level of the control group.

DETAILED DESCRIPTION:
Attention Deficit Hyperactivity disorder (ADHD) is one of the most frequent childhood disorders with an estimated prevalence of about 5%. Multimodal treatment is recommended in both national and international guidelines of ADHD care, but most patients only receive pharmacological treatment, sometimes in combination with parent training. As such, the most common treatment approach today is stimulant medication, e.g., methylphenidate. However, there are insufficient understanding about several aspects of medical treatment. For example, it is not evident that medication improves learning processes and the best dosage for cognitive functioning and adapted school behavior differs.

Original findings from our research group shows that auditory noise has the possibility of enhancing cognitive performance in inattentive children without diagnosis as well as children with an ADHD diagnosis. One study found that the benefit of noise was in parity with, or even larger than, the benefit of pharmacological ADHD treatment on two cognitive tasks. The theory about noise benefit is thoroughly described by Sikström and Söderlund (2007). If auditory or visual noise, as suggested by the present project, could be a complement, or an alternative, to stimulant medication it could fundamentally change the treatment of ADHD and the school situation for those children.

The aims of this study are to: i) evaluate the effects of auditory white noise and visual white pixel noise on cognitive performance during two eye tracking tasks, ii) compare effects between ADHD and control groups ii) link noise benefit to specific traits.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents with a diagnosis of ADHD and control children without a diagnosis

Exclusion Criteria:

* Intellectual disability
* Psychosis
* Severe depression or anxiety
* The need of an interpreter to participate in the study

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-06-01 (Actual)

PRIMARY OUTCOMES:
Inhibitory control | Six months
  Inhibitory control is the ability to suppress nonproductive behaviors and cognitive processing and will be measured through the eye tracking tasks (PF and MGS) in the study.

SECONDARY OUTCOMES:
SNAP | Six months
  The SNAP rating scale is an assessment tool for traits of hyperactivity and inattention in ADHD (Swanson et al., 2012). Will be filled out by legal guardians of the participants.
5-15R | Six months
  The 5-15R assessment is aimed at legal guardians of the participants and consists of 181 claims that evaluates motor and cognitive performance in children aged 5 to 15 as well as a psychiatric assessment (Kadesjö et al., 2017)

CONTACTS AND LOCATIONS:
Overall Officials: Emma Claesdotter-Knutsson, MD: PhD, Principal Investigator — IKVL, Lund University
Locations (1):
- Child and Adolescent Psychiatry Clinic, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Jostrup E, Nystrom M, Tallberg P, Soderlund G, Gustafsson P, Claesdotter-Knutsson E. Effects of Auditory and Visual White Noise on Oculomotor Inhibition in Children With Attention-Deficit/Hyperactivity Disorder: Protocol for a Crossover Study. JMIR Res Protoc. 2024 Aug 15;13:e56388. doi: 10.2196/56388. PMID 39146010